CLINICAL TRIAL: NCT01256645
Title: Liberal Versus Restrictive Transfusion Management in Patients Being Weaned From Prolonged Mechanical Ventilation
Brief Title: Transfusion Strategies in Weaning Patients
Acronym: WTT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Responsible Party: Koehler, Prof. Dr., Kloster Grafschaft
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WT 2010
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Weaning Patients
Keywords: weaning; mechanical ventilation; blood transfusion; spontaneous breathing trials
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- restrictive transfusion (No Intervention): No transfusion given to correct anemia unless vital indication is given
- liberal transfusion (Experimental): transfusions are given in single units until Hb is > 12 mg/dl
  Interventions: Other: blood transfusion

INTERVENTIONS:
Other: blood transfusion — application of single units of red blood cell transfusions
  Arms: liberal transfusion

SUMMARY:
The aim of this study is to determine, whether a liberal transfusion strategy is helpful to liberate patients from prolonged invasive mechanical ventilation.

Patients who are difficult to wean according to the criteria by Boles et al [1] are limited by the capacity of their respiratory muscles.

Improved oxygen delivery achieved by blood transfusions however is known to decrease the work of breathing [2] and thus in theory can improve weaning success [3].

This study is designed as a prospective, randomized, open labeled blinded End-point evaluation to test the hypothesis that a liberal transfusion strategy decreases the time needed for weaning.

1. Boles, JM, J Bion, A Connors, M Herridge, B Marsh, C Melot, R Pearl, H Silverman, M Stanchina, A Vieillard-BaronandT Welte, Weaning from mechanical ventilation. Eur Respir J, 2007. 29(5): p. 1033.
2. Schonhofer, B, M Wenzel, M GeibelandD Kohler, Blood transfusion and lung function in chronically anemic patients with severe chronic obstructive pulmonary disease. Crit Care Med, 1998. 26(11): p. 1824.
3. Schonhofer, B, H BohrerandD Kohler, Blood transfusion facilitating difficult weaning from the ventilator. Anaesthesia, 1998. 53(2): p. 181.

DETAILED DESCRIPTION:
Liberation from invasive mechanical ventilation has a huge impact on quality of life and healthcare expenses. Weaning is more difficult and complex in patients who have been ventilated for a longer time (i.e. more than seven days) or have undergone multiple failed weaning attempts and thus are classified weaning category three according to Boles at al. [1] Current national and international guidelines are in favour of a rather restrictive transfusion regime. This recommendation is mainly based on the work of Hebert et al. [2] where no benefit or a liberal transfusion approach could be found. Patients in the Hebert study however had become acutely ill and did not show any impairment or dysfunction of the respiratory muscles

Weaning class 3 patients however suffer from an overload of their respiratory muscles either cause by an increased load or decreased capacity.

In either instance unloading of the respiratory muscles is key to improve the capability of spontaneous breathing. One possible way to achieve this goal is to improve oxygen delivery.

Oxygen delivery is determined by the cardiac output times the oxygen content of the blood. The latter is mainly determined by the haemoglobin concentration and the oxygen saturation (Hb x 1.34 x SaO2 + PO2 x 0.003). Previous studies have shown that in patients with a strained respiratory pump blood transfusions improve the work of breathing [3].

A more liberal transfusion strategy therefore might improve the weaning outcome ventilator dependant patients [4]

This study is designed as a prospective, randomized, open labeled blinded End-point evaluation to test the hypothesis that a liberal transfusion strategy decreases the time needed for weaning.

Patients who are anemic (Hb < 9 mg/dl) and were admitted to our specialized weaning unit are either randomized to a conservative or liberal transfusion regime if they are agreed to participate.

The goal in the liberal transfusion group is to keep the Hb at > 12 mg/dl and transfusions are given in single units until this threshold is achieved.

Patients then undergo routine weaning procedures consistent of daily or multiple daily weaning trials paired with intermittent ventilation targeted do rest the respiratory muscles.

Daily physiologic data are recorded as well as adverse events. Primary outcome is the time needed to wean the patients off invasive mechanical ventilation, mortality is a secondary criterium.

The study is planned to include 120 patients in blocks of 40 patients. Interim analysis will be performed after each block and the study will be terminated if a significant result is achieved.

1. Boles, JM, J Bion, A Connors, M Herridge, B Marsh, C Melot, R Pearl, H Silverman, M Stanchina, A Vieillard-BaronandT Welte, Weaning from mechanical ventilation. Eur Respir J, 2007. 29(5): p. 1033.
2. Hebert, PC, G Wells, MA Blajchman, J Marshall, C Martin, G Pagliarello, M Tweeddale, I SchweitzerandE Yetisir, A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med, 1999. 340(6): p. 409.
3. Schonhofer, B, M Wenzel, M GeibelandD Kohler, Blood transfusion and lung function in chronically anemic patients with severe chronic obstructive pulmonary disease. Crit Care Med, 1998. 26(11): p. 1824.
4. Sato, T, EJ BedrickandC Tsai, Model Selection for Multivariate Regression in Small Samples. Biometrics, 1998. 54(1): p. 391.

ELIGIBILITY:
Inclusion Criteria:

* Hb < 9g/dl
* Prolonged mechanical ventilation for > 14 days
* Hemodynamically stable / no acute ongoing disease
* weainingfailure
* spontaneous breathing capacity less than four hours
* Euvolemia
* Consent

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* known blood incompatibility
* acute indications to give blood products or previous transfusions within the last three days
* previously known chronic anemia
* coma
* ongoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Time to sucessfull weaning | 14 days
  Time between randomisation an sucessfull liberation from invasive mechanical ventilation

SECONDARY OUTCOMES:
mortality | within hospital
  mortality during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Köhler, Prof, Study Chair — FKKG; Dominic Dellweg, M.D., Principal Investigator — FKKG; Thomas Barchfeld, M.D., Principal Investigator — FKKG
Locations (1):
- Kloster Grafschaft, Schmallenberg, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Schonhofer B, Bohrer H, Kohler D. Blood transfusion facilitating difficult weaning from the ventilator. Anaesthesia. 1998 Feb;53(2):181-4. doi: 10.1046/j.1365-2044.1998.00275.x. PMID 9534644
- [Background] Schonhofer B, Wenzel M, Geibel M, Kohler D. Blood transfusion and lung function in chronically anemic patients with severe chronic obstructive pulmonary disease. Crit Care Med. 1998 Nov;26(11):1824-8. doi: 10.1097/00003246-199811000-00022. PMID 9824074